CLINICAL TRIAL: NCT06711809
Title: The Role of Sleep, Oxytocin and Reward Processing in Women in the Postpartum Phase
Brief Title: Sleep, Oxytocin and Reward Processing in Women in the Postpartum Phase
Status: Not yet recruiting | Type: Observational
Sponsor: International Research Training Group 2804 (Other)
Collaborators: Uppsala University (Other); Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRTG_P06_2
Record Dates: First submitted 2024-11-22; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Postpartum Depression
Keywords: oxytocin; peripartum depression; postpartum depression; sleep; sleep assessment; reward processing; motivation
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva samples for salivary oxytocin analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
During and after pregnancy, a woman's body and brain undergo significant changes that help her adapt to caregiving and emotional needs. However, this period also makes women more susceptible to emotional disorders, such as peripartum depression (PPD), which affects about 10-15% of new mothers. PPD can negatively impact both the mother and her baby, disrupting mood, motivation, and mothering abilities. Hormonal changes and poor sleep are some of the risk factors that might worsen these depressive symptoms.

Traditionally, sleep studies on PPD have relied on questionnaires and short-term sleep assessments. With the advent of smartwatches and digital devices, we can now monitor sleep in a home environment over longer periods. Oxytocin, a hormone crucial for childbirth, breastfeeding, and bonding with the baby, is thought to play a role in PPD. Studies suggest that higher levels of oxytocin might be linked to lower levels of postpartum depression, though findings are not always consistent. Oxytocin also affects sleep and is connected to brain areas that regulate reward and motivation.

This study aims to explore the relationship between sleep, oxytocin, and reward processing in new mothers. The investigators will include women with varying levels of depressive symptoms and use home-based sleep assessments to gather data. Our goal is to better understand how these factors interact in the postpartum period and how they might influence a mother's mental health and caregiving abilities.

The investigators expect that oxytocin levels are reduced in women with higher depressive symptoms and that these reductions are associated with sleep impairments, breastfeeding and altered reward processing.

DETAILED DESCRIPTION:
The study will be conducted at Uppsala University. Data will be mainly collected at the participants' home. The investigators plan to include 100 women in the postpartum phase in total, including women with different depressive scores according to the Edinburgh Postnatal Depression Scale (EPDS). Ideally, the investigators aim to include 50 women with depressive symptoms (EPDS ≥12) and 50 women without depressive symptoms (EPDS score ≤6). However, depending on the number of available participants and recruitment efforts the investigators will possibly include all interested women in the postpartum phase to increase the feasibility of the study and use a continuous categorization of the depressive (EPDS) scores.

The participants will be asked to fill out (online) questionnaires. The investigators will assess their demographic data and socioeconomic status as well depressive symptoms (Montgommery Asberg Depression Scale (MADRS); Edinburgh Postnatal Depression Score (EPDS)) and sleep/chronotype (morningness-eveningness questionnaire (MEQ); Pittsburg Sleep Quality Index (PSQI); Ford Insomnia Response to Stress Test (FIRST); Insomnia severity index (ISI); Epworth sleepiness scale (ESS); Fatigue Severity Scale (FSS)). Additionally, the investigators will include sleep questionnaires which are specific for the postpartum phase (Postpartum Sleep Quality Scale (PSQS)) and ask the mothers to rate the infants sleep using the Brief Infant Sleep Questionnaire (BISQ-R). Participants will be asked to fill out questionnaire regarding their breastfeeding behavior (Breastfeeding Self-Efficacy Scale Short Form (BSES-SF); Baby Eating Behavior Questionnaire (BEBQ)), bonding (Postpartum Bonding Questionnaire (PBQ); Swedish mother to infant bonding scale (S-MIBS)) and reward processing (indecisiveness scale IS, action regulation ARES).

Participants will take part in an online behavioral task ("Effort Allocation Task (EAT)") that assesses reward processing, in particular motivation for primary rewards (i.e. food) and secondary rewards (i.e. money) (approximately 20 minutes).

The experimenter will explain all the procedures for the at-home assessment and participants will be given the devices accordingly. For the at-home measurement of sleep, participants will receive tracking devices (Fitbit Inspire; Withings sleep analyser) which they should use for one week (7 days) to assess sleep multimodally. The Fitbit will also assess daily physiological measures i.e., physical activity during the day and heart rate. Additionally, subjective sleep, breastfeeding and the current mood will be assessed at several timepoints throughout the week using standardized diaries and questionnaires.

Furthermore, the participants will receive saliva sample kits to use at different timepoints throughout the measurement period to assess endogenous oxytocin levels. If participants are breastfeeding, the investigators will additionally ask them to take saliva samples before and after a breastfeeding period to assess changes in salivary oxytocin associated with breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Biological sex/gender: female
* Swedish/English fluency
* Postpartum phase: 6 weeks to 1 year

Exclusion Criteria:

* Age < 18
* Neonatal complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Research participants will be recruited in the area of Uppsala, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
objective sleep | 7 consecutive nights
  Objective sleep measures assessed with tracking devices (Fitbit Inspire; Withings sleep analyser) e.g., total time spent in bed, wake time, wake frequency, sleep stages duration.
subjective sleep | 7 consecutive days
  Subjective sleep assessed by a daily sleep diary.
oxytocin levels | 7 consecutive days
  Oxytocin levels assessed with saliva kits.
breastfeeding | 7 consecutive days
  Assessment of breastfeeding behavior (onset, frequency and duration) with breastfeeding diaries.
bonding | 7 consecutive days
  Bonding of mother and child assessed with questionnaires.
reward processing/motivation | 7 consecutive days
  Assessment of effort-based motivation using the effort allocation task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Uppsala, Uppsala, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: Undecided